CLINICAL TRIAL: NCT06406075
Title: A Pilot Study to Assess the Ability of Advanced Spectroscopy Techniques and Machine Learning Models to Non-invasively Measure Glucose Robustly and Accurately
Brief Title: Non-invasive Measurement of Glucose with Advanced Spectroscopy Techniques and Machine Learning Models
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liom Health AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPN-006
Record Dates: First submitted 2024-04-11; First posted 2024-05-09 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Continuous glucose monitoring; Noninvasive; Transcutaneous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational arm (Experimental): Induction of glycose dynamics and collection of transcutaneous spectral data and reference glucose values
  Interventions: Device: Lab demo 1.0

INTERVENTIONS:
Device: Lab demo 1.0 — During the intervention, transcutaneous spectral data are collected continuously with the Lab demo. Up to 20 whole blood glucose reference values are also collected, as well as interstitial fluid glucose values using a continuous glucose monitoring device. Some participants will attend multiple measurement sessions.

SUMMARY:
Primary aim of this pilot study is to provide evidence for a non-invasive, continuous, and transcutaneous measurement method to determine blood glucose levels robustly and accurately.

DETAILED DESCRIPTION:
The study is divided into 3 sub-studies focusing on

* Interchangeability of Lab demo 1.0
* Evaluation of advanced spectroscopy methods and their miniaturisation potential
* Robustness of machine learning model to changes over time

ELIGIBILITY:
Inclusion Criteria:

* Provide signed and dated written informed consent by study participant prior to any mandatory study-specific procedures, sample collection, or analysis
* Apparently healthy Male or Female adult aged between 18 and 75
* Willingness to follow the study procedures

Exclusion Criteria:

* In Female subjects: pregnancy or breastfeeding period
* A diagnosis of diabetes mellitus (any type) with ongoing insulin therapy (basal or basal plus bolus) or sulfonylurea therapy
* Prior severe hypoglycemia event (stage 3 or above; e.g., seizure, loss of consciousness, emergency hospitalisation)
* Prior event of severe hyperglycemia resulting in diabetic ketoacidosis or hyperosmolar hyperglycemic state, or emergency hospitalisation
* Documented medical history of bleeding disorder
* Being under anticoagulant medication
* Insufficient knowledge of project languages (English/German)
* Known sensitivity to medical-grade adhesives or other skin-related complications, which might influence the outcome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Comparison of glucose changes measured over a time series of transcutaneous measurements with reference measurements | The data is collected during the study procedure (up to 3 hours)
  The transcutaneous glucose measurements and the corresponding spectral fingerprints are compared with the values of interstitial fluid (ISF) and capillary blood glucose.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien Rebeaud, PhD, Study Director — Liom Health AG
Locations (1):
- Liom Health AG, Pfaeffikon, Canton of Schwyz, Switzerland

IPD SHARING:
Plan to Share IPD: No